CLINICAL TRIAL: NCT06469476
Title: Evaluation of Access to Screening for Post-partum Depression Via the Postnatal Interview Within 8 Weeks of Birth in Women Who Have Gave Birth at the Troyes Hospital ( DEPRESSIONPP )
Acronym: DEPRESSIONPP
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Troyes (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02394-41
Record Dates: First submitted 2024-05-31; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Depression, Postpartum
Keywords: depression post partum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: depression post partum — visit post partum

SUMMARY:
Post-partum depression is defined as a depressive disorder with onset of symptoms in the year following childbirth. Several international studies have reported a prevalence of this condition of around pathology of around 15%. Santé publique France's 2021 national perinatal survey corroborated these figures, finding a prevalence of post-partum depression in France of in France of 16.7%. It is therefore a frequent pathology that can cause complications for both mother and child.

The complications both for the mother and for the mother-child bond. Indeed, post-partum depression can lead to an increased risk of infanticide, weaker mother-child attachment, and altered parental behaviour. post-partum depression can lead to maternal suicide (the second leading cause cause of maternal mortality in France). Despite the potential seriousness of severe depression and its impact on the on the mother-child bond, just under half of those suffering from severe depression suffering from severe depression consult a healthcare professional.

Fear of being judged or stigmatised, linked to misperceptions about the episode, is one of the main obstacles to consultation.

Of being judged or stigmatised, linked to erroneous representations of the depressive episode. Given the scale of this condition, and the difficulties young mothers face in seeking help for young mothers to seek help, it is vital to screen postpartum women as widely and post-partum women as early as possible. In view of the extent of this condition and the difficulties young mothers have in seeking help for young mothers, it is vital to screen post-partum women as widely and as post-partum. With this in mind, from July 2022, a compulsory early post-natal interview has been introduced, designed to screen for postpartum depression.

DETAILED DESCRIPTION:
Main objective: To evaluate the associated factors, in particular referral by a professional as a determinant of whether or not the 'compulsory' early interview.

Secondary objective: To assess the economic, geographical and other factors associated and other factors associated with the compulsory early postnatal interview. Type of study: Observational, retrospective study. Population: Women who gave birth at the Centre Hospitalier de Troyes from July 2022 to October 2023. Assessment criteria : To be referred or not by a health professional during the early postnatal interview. Investigation plan: Send the information note and no objection to all eligible eligible women, together with the questionnaire and a T envelope to return the completed questionnaire. Inclusion criteria The study will include adult women who have given birth at the Centre hospitalier de Troyes between July 2022 and October 2023 and agreeing to take part in the study. Non-inclusion criteria The following will not be included in the study

* minors under the age of 18
* those protected by law (guardianship, curatorship and safeguard of justice)
* patients refusing to participate in the study

ELIGIBILITY:
Inclusion criteria:

* The study will include adult women who have given birth at the Centre hospitalier de Troyes from July 2022 to October 2023
* and agreeing to take part in the study.

non inclusion criteria

* minors under the age of 18
* those protected by law (guardianship, curatorship and safeguard of justice)
* patients refusing to take part in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: the adult women who have given birth at the Centre Hospitalier de Troyes between July 2022 and October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Measure if the patient is yes or not to be referred by a healthcare professional during the early postnatal interview. | 3 months
  question

SECONDARY OUTCOMES:
Measure the socio-economic status | 3 months
  financial parameter
measure the declaration of a financial or non-financial obstacle | 3 months
  financial parameter
measure the knowledge about post-partum depression | 3 months
  question first contact
measure the knowledge about early post-natal interview. | 3 months
  question

CONTACTS AND LOCATIONS:
Overall Officials: Amjad KATTINI, DR, Principal Investigator — Centre Hospitalier de Troyes
Locations (1):
- Centre Hospitalier de Troyes, Troyes, Grand Est, France

IPD SHARING:
Plan to Share IPD: Undecided